CLINICAL TRIAL: NCT02657044
Title: Multicenter, Randomised Controlled Trial Comparing Endoscopic Mucosal Resection (EMR) And Endoscopic Submucosal dissecTIon (ESD) for Resection of Large Distal Non-pedunculated Colorectal Adenomas (MATILDA-trial)
Brief Title: EMR Versus ESD for Resection of Large Distal Non-pedunculated Colorectal Adenomas
Acronym: MATILDA
Status: Unknown | Phase: Not Applicable | Type: Interventional
Last Known Status: Recruiting
Sponsor: UMC Utrecht (Other)
Collaborators: Comprehensive Cancer Centre The Netherlands (Other)
Responsible Party: Principal Investigator, L.M.G. Moons, dr. L.M.G. Moons, Principal Investigator, UMC Utrecht
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: 15-610/D; TDM-H1/8051 (Other Grant/Funding Number: Dutch Cancer Society (DCS))
Record Dates: First submitted 2016-01-08; First posted 2016-01-15 (Estimated); Last update posted 2016-10-26 (Estimated); Status verified 2016-10

CONDITIONS: Colorectal Neoplasms
Keywords: EMR; ESD; endoscopic mucosal resection; endoscopic submucosal resection; colorectal adenomas
MeSH Terms: conditions — Colorectal Neoplasms | interventions — Endoscopic Mucosal Resection

STUDY DESIGN:
Oversight: Data Monitoring Committee: No

ARMS (2):
- EMR (Active Comparator): In the EMR-arm, endoscopic resection will be performed using the (p)EMR technique.
  Interventions: Procedure: EMR
- ESD (Active Comparator): In the ESD-arm, endoscopic resection will be performed using the (h)ESD technique.
  Interventions: Procedure: ESD

INTERVENTIONS:
Procedure: EMR
  Other Names: Endoscopic Mucosal Resection
  Arms: EMR
Procedure: ESD
  Other Names: Endoscopic Submucosal Dissection
  Arms: ESD

SUMMARY:
Endoscopic resection of adenomas in the colon is the cornerstone of effective colorectal cancer prevention. Endoscopic mucosal resection (EMR) is currently the most used technique for resection of large distal colorectal adenomas, however, maintains some important limitations. In large lesions, EMR can often only be performed in a piecemeal fashion resulting in relatively low R0-resection rates and high recurrence rates. Endoscopic submucosal dissection (ESD) is a newer procedure that is more difficult resulting in a longer procedural time, but is promising due to the high en-bloc resection rates and the very low recurrence rates. The aim of this multicenter randomized study is to compare EMR and ESD with regard to recurrence rates and radical (R0) resection rates, and to put this into perspective against the costs and complication rates of both strategies and the burden perceived by patients on the long term-term.

ELIGIBILITY:
Inclusion Criteria:

* non-pedunculated polyp larger than 20 mm in the rectum, sigmoid or descending colon found during colonoscopy
* indication for endoscopic treatment
* ≥18 years old
* Written informed consent

Exclusion Criteria:

* suspicion of malignancy, as determined by endoscopic findings (invasive Kudo pit pattern, Hiroshima type C) or proven malignancy at histology
* prior endoscopic resection attempt
* presence of synchronous distal advanced carcinoma that requires surgical resection
* the risk exceeds the benefit of endoscopic treatment, such as patient's with an extremely poor general condition or a very short life expectancy
* the inability to provide informed consent

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 212 (Estimated)
Dates: Start 2016-04; Primary Completion 2018-09 (Estimated); Study Completion 2020-12 (Estimated)

PRIMARY OUTCOMES:
Recurrence rate at follow-up colonoscopy after 6 months | 6 months
  Observed from resected residual disease or, if not present, from biopsies of the scar

SECONDARY OUTCOMES:
Long-term recurrence rate at follow-up colonoscopy after 36 months | 36 months
  Observed from resected residual disease or, if not present, from biopsies of the scar
Health care resource utilization and consts | 36 months
  Healthcare costs will be calculated by multiplying used healthcare services with unit prices. The cost-effectiveness of ESD against EMR will be expressed as incremental cost-effectiveness ratios (ICER) showing additional costs per recurrence free patient and as ICER showing additional costs per QALY.
Perceived burden and quality of life among patients | 36 months
  Measurement of the patients' burden of ESD versus EMR will be evaluated with regard to colorectal cancer anxiety, burden of the procedure itself, functional complaints and overall quality of life. Meaurement will be performed using validated questionnaires.
Complication rate | 30 days
  Complications will be assessed on day 30: intraprocedural perforation, Intraprocedural bleeding, Postprocedural bleeding, Postprocedural perforation, Postprocedural serositis.
Surgical referral rate | 36 months
  Defined as the number of patients that are referred for surgical management at 36 months
R0-resection rate | 30 days
  Defined as dysplasia free vertical and lateral resection margins at histology

CONTACTS AND LOCATIONS:
Overall Officials: L.M.G. Moons, MD, PhD, Principal Investigator — UMC Utrecht; A.D. Koch, MD, PhD, Principal Investigator — Erasmus Medical Center
Locations (1):
- UMC Utrecht, Utrecht, Utrecht, Netherlands

REFERENCES:
- [Derived] Backes Y, Moons LM, van Bergeijk JD, Berk L, Ter Borg F, Ter Borg PC, Elias SG, Geesing JM, Groen JN, Hadithi M, Hardwick JC, Kerkhof M, Mangen MJ, Straathof JW, Schroder R, Schwartz MP, Spanier BW, de Vos Tot Nederveen Cappel WH, Wolfhagen FH, Koch AD. Endoscopic mucosal resection (EMR) versus endoscopic submucosal dissection (ESD) for resection of large distal non-pedunculated colorectal adenomas (MATILDA-trial): rationale and design of a multicenter randomized clinical trial. BMC Gastroenterol. 2016 May 26;16(1):56. doi: 10.1186/s12876-016-0468-6. PMID 27229709